CLINICAL TRIAL: NCT06086938
Title: Personalized Brain Functional Sector-guided Continuous Theta Burst Stimulation Combined With Intermittent Theta Burst Stimulation Therapy Targeting at the Superior Frontal Gyrus for Aphasia After Ischemic Stroke: a RCT
Brief Title: pBFS-guided cTBS Combined With iTBS Over the Superior Frontal Gyrus for Aphasia After Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changping Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPSA07BJ40
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Stroke, Ischemic; Aphasia
MeSH Terms: conditions — Ischemic Stroke; Aphasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active TBS group (Active Comparator): active TBS combined with speech language therapy
  Interventions: Device: active cTBS combined with iTBS
- sham TBS group (Sham Comparator): sham TBS combined with speech language therapy
  Interventions: Device: sham cTBS combined with iTBS

INTERVENTIONS:
Device: active cTBS combined with iTBS — Daily TBS treatment consists of the following combination: active 600-pulse cTBS applied to the superior frontal gyrus (SFG) in the unaffected hemisphere + active 600-pulse iTBS applied to the SFG in the affected hemisphere + 15 minutes of rest + active 600-pulse cTBS applied to the SFG in the unaffected hemisphere + active 600-pulses iTBS applied to the SFG in the affected hemisphere, totaling 2400 pulses of TBS intervention.
  The intervention mentioned above will be administered once per day with five consecutive days per week, continuously for three weeks.
  Arms: active TBS group
Device: sham cTBS combined with iTBS — Daily sham TBS treatment consists of the following combination: sham 600-pulse cTBS applied to the superior frontal gyrus (SFG) in the unaffected hemisphere + sham 600-pulse iTBS applied to the SFG in the affected hemisphere + 15 minutes of rest + sham 600-pulse cTBS applied to the SFG in the unaffected hemisphere + 600-pulse sham iTBS applied to the SFG in the affected hemisphere, totaling 2400 pulses of sham TBS intervention.
  The intervention mentioned above will be administered once per day with five consecutive days per week, continuously for three weeks.
  Arms: sham TBS group

SUMMARY:
The current study aims to evaluate the efficacy and safety of pBFS-guided cTBS combined with iTBS for the rehabilitation of language functions in patients with post-ischemic stroke aphasia.

DETAILED DESCRIPTION:
Increasing evidence suggests that rTMS has been effective in treating various psychological and neurological diseases, including treating post-stroke symptoms. Using the personalized brain functional sectors (pBFS) technique, we could precisely identify individualized brain functional networks and the personalized language-related stimulation site based on the resting-state functional MRI data. The current study proposes to conduct a double-blinded, randomized and parallel controlled design trial, to investigate the efficacy and safety of pBFS-guided personalized cTBS combined with iTBS intervention in post-stroke aphasic patients.

Subjects will be randomly assigned to the following two groups: active TBS（cTBS+iTBS）group, or a sham TBS（sham cTBS+sham iTBS）group. The allocation ratio will be 1:1. The stimulation protocol consisted of a 3-week treatment, with five consecutive days each week (totally 15 day-treatment) .The stimulation procedure will be assisted with real-time neuronavigation to ensure its precision.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's age ranges from 35 to 75 years old (including 35 and 75 years old);
2. Meet the diagnostic criteria for acute ischemic stroke (diagnosed according to the "Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke" written by the American Heart Association/American Stroke Association in 2019 and the "Chinese Guidelines for Diagnosis and Treatment of Acute Ischemic Stroke 2018" compiled by the Neurology Branch of the Chinese Medical Association in 2018), with lesions in the left hemisphere, and a duration of ≥15 days and ≤3 months;
3. Diagnosed as aphasia patient according to the Chinese version of Western Aphasia Battery (WAB), with a WAB-aphasia quotient of less than 93.8 points;
4. First onset of stroke;
5. Normal functioning language abilities before the stroke, with Mandarin as their native language and an educational level higher than primary school；
6. Understand the trial and signed the informed consent form.

Exclusion Criteria:

1. Combined severe dysarthria (NIHSS item 10 score ≥2 points);
2. Aphasia caused by bilateral hemisphere stroke, brain tumor, traumatic brain injury, Parkinson's disease, motor neuron disease, or other diseases；
3. Patients with implanted electronic devices such as cardiac pacemakers, cochlear implants, or other metal foreign bodies, or those with MRI contraindications such as claustrophobia or TMS treatment contraindications;
4. History of epilepsy;
5. Patient with concomitant severe systemic diseases affecting the heart, lungs, liver, kidneys, etc., and uncontrolled by conventional medication, as detected and confirmed through laboratory testing and examination;
6. Patients with consciousness disorders (NIHSS 1(a) score ≥1);
7. Patients with malignant hypertension;
8. Patients with severe organic diseases, such as malignant tumors, with an expected survival time of less than 1 year;
9. Patients with severe hearing, visual, cognitive impairment or inability to cooperate with the trial;
10. Patients with severe depression, anxiety, or diagnosed with other mental illnesses that prevent them from completing the trial;
11. Patients who have received other neuroregulatory treatments such as TMS, transcranial electric stimulation, etc. in the 3 months prior to enrollment;
12. Patients with a history of alcoholism, drug abuse, or other substance abuse;
13. Patients with other abnormal findings that the researchers judge are not suitable for participation in this trial;
14. Patients who are unable to complete follow-up due to geographical or other reasons;
15. Women of childbearing age who are currently pregnant, breastfeeding, or planning or may become pregnant during the trial;
16. Patients who are currently participating in other clinical trials.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Change in the Western Aphasia Battery scores | baseline, end of the 3-week therapy
  The first four subsets of the WAB (Spontaneous Speech, Auditory verbal comprehension, Repetition, Naming and word finding) will be used to evaluate the participants' language ability impairments. A Chinese adapted version of WAB will be used. The scores from all four subsets will be calculated as an Aphasia Quotient (ranging from 0 to 100), with lower Aphasia Quotients indicating poorer language abilities.

SECONDARY OUTCOMES:
Change in the Western Aphasia Battery scores | baseline, end of the 5-day therapy, 90 days after treatment initiation
  The first four subsets of the WAB (Spontaneous Speech, Auditory verbal comprehension, Repetition, Naming and word finding) will be used to evaluate the participants' language ability impairments. A Chinese adapted version of WAB will be used. The scores from all four subsets will be calculated as an Aphasia Quotient (ranging from 0 to 100), with lower Aphasia Quotients indicating poorer language abilities.
Boston Diagnostic Aphasia Examination Severity Ratings | baseline，end of the 3-week therapy，90 days after treatment initiation
  The Boston Diagnostic Aphasia Examination (BDAE) Severity Ratings is a clinical tool used to evaluate the severity and type of aphasia in individuals. The assessment includes four domains: communication abilities, language content, speech sound production and response abilities.BDAE severity ratings range from level 0 to level 5, with lower scores indicating more severe aphasia.
Chinese-version Stroke and Aphasia Quality of Life Scale 39-generic version (SAQOL-39g) | baseline，end of the 3-week therapy，90 days after treatment initiation
  The SAQOL-39g is a quality of life assessment tool that is used to evaluate the impact of stroke and aphasia on a patient's quality of life. It consists of 39 items that cover a range of domains related to the patient's quality of life, such as communication, physical functioning, mood, and social support. The items are rated on a 5-point Likert scale ranging from "not at all" to "very much", with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory